CLINICAL TRIAL: NCT03395236
Title: ProspectIve, MuLti-Center Study to EvaLUate TreatMent of Subjects With OcclusivE Disease With a Novel PAcliTazel-CoatEd Angioplasty Balloon in Below-The-Knee (BTK) Arteries: a Post Market Clinical Study
Brief Title: ILLUMENATE Below-The-Knee (BTK) Arteries: a Post Market Clinical Study
Acronym: BTK PMS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Spectranetics Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D037012
Record Dates: First submitted 2017-12-01; First posted 2018-01-10 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2023-11

CONDITIONS: Peripheral Arterial Disease
Keywords: Critical Limb Ischemia; CLI; Claudication; PAD; BTK; Below The Knee
MeSH Terms: conditions — Peripheral Arterial Disease; Chronic Limb-Threatening Ischemia; Intermittent Claudication

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Treatment (Experimental): StellarexTM 0.014 OTW Drug-coated Angioplasty Balloon (Stellarex Balloon)
  Interventions: Combination Product: StellarexTM 0.014" Over-The-Wire Drug-coated Angioplasty Balloon

INTERVENTIONS:
Combination Product: StellarexTM 0.014" Over-The-Wire Drug-coated Angioplasty Balloon — The Stellarex balloon (0.014") is indicated for the treatment of de-novo or re-stenotic lesions in the lower extremities to establish blood flow and to maintain vessel patency.

SUMMARY:
The objective of this prospective, multi-center, single arm study is to obtain further data on the safety and performance of the StellarexTM 0.014" OTW Drug-coated Angioplasty Balloon in the treatment of lesions in "below the knee" popliteal (P3 segment) and infra-popliteal arteries according to the Instructions for Use in Rutherford-Becker Classification (RCC) 3, 4 and 5 patient populations. This study will be conducted in Europe across up to 10 centers in up to 75 subjects. Office visits will occur at 30 days, 6, 12, and 24 months post-index procedure.

DETAILED DESCRIPTION:
There is a significant amount of evidence that the use of Paclitaxel-coated balloons in the treatment of peripheral arterial disease (PAD) has demonstrated favorable outcomes when used to treat lesions in the superficial femoral and popliteal arteries. For subjects with lesions in the infrapopliteal arteries, which includes lesions in the mid to distal popliteal artery and below, a smaller profile balloon is necessary. Typically, lesions in the SFA and proximal popliteal arteries are treated by larger diameter balloons and larger sized guidewires (most commonly 0.018" or 0.035") which are too large for vessels below-the-knee. For this reason, the Stellarex™ 0.014" OTW Drug-coated Angioplasty Balloon was developed as a line extension to the Stellarex™ 0.035" device in order to accommodate the treatment of these smaller vessels. The Stellarex™ 0.014" balloon has the same drug concentration and is manufactured using a similar method as the Stellarex™ 0.035" device. Additionally, the Stellarex™ 0.035" and 0.014" balloon share a common balloon diameter of 4 mm, a size which was used to treat lesions throughout the popliteal artery in the previous Stellarex 0.035" studies. For the reasons noted above, equivalence between the two devices has been demonstrated. Furthermore, it is believed that the 0.014" device will not demonstrate any performance differences nor change the anticipated or residual risks.

In conclusion, the current study has been developed in agreement with post-market requirements as per the Post Market Clinical Follow up (PMCF) plan. The prospective design of the study, the sample size and the selected outcomes will be able to provide the additional clinical information to support the safe use and performance of the Stellarex 0.014" device in the intended population of patients with below-the-knee arterial disease.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects intended to be treated with the Stellarex 0.014" Drug-Coated Balloon for de-novo or restenotic lesions in native "below the knee" popliteal (P3 segment) and infra-popliteal arteries ending at the tibiotalar joint (ankle), as per the Instruction for Use (IFU).
2. Rutherford-Becker clinical category classification (RCC) 3 patients with claudication or RCC 4 or 5 subjects with documented Critical Limb Ischemia (CLI) defined as 2.1 RCC 3 subjects: subjects with severe claudication 2.2 RCC 4 subjects: subjects with persistent, recurring ischemic rest pain requiring analgesia for at least two weeks or 2.3 RCC 5 subjects: subjects with minor tissue loss of the foot or toes or
3. Age ≥18 years old.
4. Reconstitution of the target vessel at the ankle and run-off into a patent dorsalis pedis or plantar arteries defined as <50% stenosis by visual estimate.
5. Is able and willing to provide written informed consent and comply with all required follow-up evaluations within the defined follow-up visit windows prior to enrollment in the study.
6. Life expectancy > 1 year.

Exclusion Criteria:

1. Subjects with any medical condition that would make him/her inappropriate for treatment with the Stellarex balloon as per the Instructions for Use (IFU) or in the opinion of the investigator.
2. Has impaired renal function defined as serum creatinine >2.5 mg/dl that cannot be adequately pre-treated or subjects on dialysis.
3. Subjects already enrolled in other investigational (interventional) studies that would interfere with study endpoints.
4. Subjects that in the judgment of the investigator would require treatment of the contralateral limb within 3 days prior to the index procedure or 30 days after. Note: Unless contralateral treatment is required to facilitate adequate access to the target lesion (e.g. contralateral iliac).
5. Previous or planned surgical or catheter-based procedure within 3 days before or 30 days after the index procedure. Note: This excludes successful inflow artery treatment within the same hospitalization or a documented preplanned minor amputation.

   * Successful inflow artery treatment is defined as attainment of residual diameter stenosis ≤ 30% without major vascular complication (e.g. absence of flow-limiting dissection, embolic event). These inflow arteries must be treated without the need for laser, atherectomy, thrombectomy, cryoplasty, brachytherapy and cutting/scoring balloons. Treatment with a Stellarex DCB of the inflow lesion, if according to its intended use, is allowed.
6. Prior endovascular treatment of the target lesion within three (3) months of the index procedure.
7. Prior stent placement in the target lesion(s).
8. Single focal lesion < 4cm in length in the absence of additional treatable popliteal or infra-popliteal lesions.
9. Subjects confined to bed that are completely non-ambulatory.
10. For RCC 5 subjects: Non-arterial ulcers such as venous ulcers, neurotrophic ulcers, heel pressure ulcers, ulcers potentially involving calcaneus region or ulcers in the proximal one-half of the foot or higher (from mid-foot and higher going up the leg).
11. Subjects scheduled to undergo a planned major amputation.
12. Presence of concentric calcification that precludes adequate vessel preparation per IFU.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2018-04-20 (Actual); Primary Completion 2023-08-23 (Actual); Study Completion 2023-08-23 (Actual)

PRIMARY OUTCOMES:
Primary Safety Endpoint-Composite Major Adverse Limb Events (MALE) + perioperative death (POD); the composite is the number of participants who do not have MALE or POD at 30 days | 30 days
  Major Adverse Limb Event (MALE) is defined as the composite of either major amputation or major re-intervention through 30 days of the index procedure. Major re-intervention is defined as creation of a new surgical bypass graft, the use of thrombectomy or thrombolysis or a major surgical graft revision such as a jump graft or an interposition graft. This is a single endpoint as it is a composite only subjects who do not have MALE or POD will be counted toward this endpoint MALE is defined as the composite of either major amputation or major re-intervention through 30 days of the index procedure. Major re-intervention is defined as creation of a new surgical bypass graft, the use of thrombectomy or thrombolysis or a major surgical graft revision such as a jump graft or an interposition graft. POD is all-cause death through 30 days of the index procedure.
Primary Performance Endpoint-Composite patency + limb salvage through 6 months; the composite is the number of participants with patency and limb salvage at 6 months | 6 months
  Patency defined as freedom from occluded target lesions (flow/no flow) verified by duplex ultrasound and clinically-driven target lesion revascularization (CD-TLR) Freedom from major amputation in the Target Limb
  This is a single endpoint as only subjects with both patency and limb salvage will be considered for this endpoint.

SECONDARY OUTCOMES:
Major adverse event (MAE) rate at 6,12, and 24 months post index procedure | 6 Months
  Defined as a composite rate of all-cause death, target limb major amputation and CD-TLR
Major adverse event (MAE) rate at 6,12, and 24 months post index procedure | 12 months
  Defined as a composite rate of all-cause death, target limb major amputation and CD-TLR
Major adverse event (MAE) rate at 6,12, and 24 months post index procedure | 24 months
  Defined as a composite rate of all-cause death, target limb major amputation and CD-TLR
Rate of CD-TLR at 6, 12 and 24 months | 6 months
  Rate of CD-TLR
Rate of CD-TLR at 6, 12 and 24 months | 12 months
  Rate of CD-TLR
Rate of CD-TLR at 6, 12 and 24 months | 24 months
  Rate of CD-TLR
Patency rate at 6, 12 and 24 months, defined as the presence of target lesion flow (absence of occlusion or no flow) as determined by Duplex Ultrasound (DUS) and freedom from CD-TLR | 6 months
  Patency rate
Patency rate at 6, 12 and 24 months, defined as the presence of target lesion flow (absence of occlusion or no flow) as determined by Duplex Ultrasound (DUS) and freedom from CD-TLR | 12 months
  Patency rate
Patency rate at 6, 12 and 24 months, defined as the presence of target lesion flow (absence of occlusion or no flow) as determined by Duplex Ultrasound (DUS) and freedom from CD-TLR | 24 months
  Patency rate
Rate of procedural complications defined as occurrence of all-cause death, stroke, myocardial infarction, emergent surgical revascularization, significant distal embolization in target limb, or thrombosis of target vessel through the end of the procedure | through study completion, approximately 5 years
  Rate of procedural complications
Rate of device or procedure related death at 30 days | 30 days
  Rate of device or procedure related death
Rate of major target limb amputation at 6 months post-procedure | 6 months
  Rate of major target limb amputation
Rate of major target limb amputation at 12 months post-procedure | 12 months
  Rate of major target limb amputation
Rate of major target limb amputation at 24 months post-procedure | 24 months
  Rate of major target limb amputation
Rate of clinically driven target vessel revascularization through 6 months | 6 months
  Rate of clinically driven target vessel revascularization
Rate of clinically driven target vessel revascularization through 12 months | 12 months
  Rate of clinically driven target vessel revascularization
Rate of clinically driven target vessel revascularization through 24 months | 24 months
  Rate of clinically driven target vessel revascularization
Lesion success: | Through study completion, approximately 5 years
  Achievement of a final in-lesion residual diameter stenosis of <50% (as determined by the angiographic core laboratory), using allowed pretreatment devices after guidewire passage through the lesion
Technical success: | Through study completion, approximately 5 years
  Achievement of a final in-lesion residual diameter stenosis of <50% (as determined by the angiographic core laboratory), using the Stellarex 0.014" Drug-Coated Balloon without a device malfunction after a guidewire passage through the l
Change in waveforms/TcPO2 from pre-procedure to 30 days | 30 days
  Change in waveforms/TcPO2 from pre-procedure
Change in waveforms/TcPO2 from pre-procedure to 6 months | 6 months
  Change in waveforms/TcPO2 from pre-procedure
Change in waveforms/TcPO2 from pre-procedure to 12 months | 12 months
  Change in waveforms/TcPO2 from pre-procedure
Change in waveforms/TcPO2 from pre-procedure to 24 months | 24 months
  Change in waveforms/TcPO2 from pre-procedure
Change in ankle-brachial index (ABI) from pre-procedure to 30 days | 30 days
  Change in ankle-brachial index (ABI) from pre-procedure
Change in ankle-brachial index (ABI) from pre-procedure to 6 months | 6 months
  Change in ankle-brachial index (ABI) from pre-procedure
Change in ankle-brachial index (ABI) from pre-procedure to 12 months | 12 months
  Change in ankle-brachial index (ABI) from pre-procedure
Change in ankle-brachial index (ABI) from pre-procedure to 24 months | 24 months
  Change in ankle-brachial index (ABI) from pre-procedure
Change in toe pressures (TP) from pre-procedure to 30 days | 30 days
  Change in toe pressures (TP) from pre-procedure
Change in toe pressures (TP) from pre-procedure to 6 months | 6 months
  Change in toe pressures (TP) from pre-procedure
Change in toe pressures (TP) from pre-procedure to 12 months | 12 months
  Change in toe pressures (TP) from pre-procedure
Change in toe pressures (TP) from pre-procedure to 24 months | 24 months
  Change in toe pressures (TP) from pre-procedure
Change in Rutherford-Becker Classification (RCC) from pre-procedure to 30 days | 30 days
  Change in Rutherford-Becker Classification (RCC) from pre-procedure
Change in Rutherford-Becker Classification (RCC) from pre-procedure to 6 months | 6 months
  Change in Rutherford-Becker Classification (RCC) from pre-procedure
Change in Rutherford-Becker Classification (RCC) from pre-procedure to 12 months | 12 months
  Change in Rutherford-Becker Classification (RCC) from pre-procedure
Change in Rutherford-Becker Classification (RCC) from pre-procedure to 24 months | 24 months
  Change in Rutherford-Becker Classification (RCC) from pre-procedure
Change in EQ-5D from pre-procedure to 30 days | 30 days
  Change in EQ-5D-5L (EuroQual-5 Dimension scale set and Visual Analog Scale score) from pre-procedure. Dimension score reporting will be determined at time of reporting and VAS score will be reported based on subject indicated scale from 0 to 100, where higher scores indicate positive outcome improvement.
Change in EQ-5D from pre-procedure to 6 months | 6 months
  Change in EQ-5D-5L (EuroQual-5 Dimension scale set and Visual Analog Scale score) from pre-procedure. Dimension score reporting will be determined at time of reporting and VAS score will be reported based on subject indicated scale from 0 to 100, where higher scores indicate positive outcome improvement.
Change in EQ-5D from pre-procedure to 12 months | 12 months
  Change in EQ-5D-5L (EuroQual-5 Dimension scale set and Visual Analog Scale score) from pre-procedure. Dimension score reporting will be determined at time of reporting and VAS score will be reported based on subject indicated scale from 0 to 100, where higher scores indicate positive outcome improvement.
Change in EQ-5D from pre-procedure to 24 months | 24 months
  Change in EQ-5D-5L (EuroQual-5 Dimension scale set and Visual Analog Scale score) from pre-procedure. Dimension score reporting will be determined at time of reporting and VAS score will be reported based on subject indicated scale from 0 to 100, where higher scores indicate positive outcome improvement.
In RCC 5 subjects, percentage of wounds healed from baseline to 30 days post-procedure as reported by the Investigator at the Investigative site | 30 days
  In RCC 5 subjects, percentage of wounds healed from baseline
In RCC 5 subjects, percentage of wounds healed from baseline to 6 months post-procedure as reported by the Investigator at the Investigative site | 6 months
  In RCC 5 subjects, percentage of wounds healed from baseline
In RCC 5 subjects, percentage of wounds healed from baseline to 12 months post-procedure as reported by the Investigator at the Investigative site | 12 months
  In RCC 5 subjects, percentage of wounds healed from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar Tepe, MD, Principal Investigator — Institut für Diagnostische und Interventionelle Radiologie, RoMed Klinikum Rosenheim
Locations (10):
- Germany (5):
  - Cardiologisches Centrum Bethanien, Frankfurt
  - Asklepios Kliniken Hamburg GmbH, Hamburg
  - Klinik Immenstadt, Herz und GefaSzentrum Immenstadt, Immenstadt im Allgäu
  - Universitatsmedizin der Johannes Gutenberg-Universitat Mainz, Mainz
  - RoMed Klinikum Rosenheim, Rosenheim
- Netherlands (2):
  - Albert Schweitzer Hospital, Dordrecht
  - St. Antonius Hospital, Nieuwegein
- United Kingdom (3):
  - Cambridge University Hospital, Cambridge
  - Guys and St. Thomas Hospital, London
  - The Royal Free Hospital, London

IPD SHARING:
Plan to Share IPD: No